CLINICAL TRIAL: NCT07017270
Title: Glucagon-like-peptide-1 Receptor Agonists in Patients Receiving Maintenance Dialysis
Acronym: GUARD-1
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO5185
Record Dates: First submitted 2025-04-24; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Kidney Disease, Chronic; Diabetes; Dialysis; End Stage Kidney Disease (ESRD)
Keywords: Dialysis; Type 2 diabetes; semaglutide; end stage kidney disease; GLP1; GLP1RA
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Kidney Failure, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): This treatment arm comprises a strategy of usual care for type 2 diabetes mellitus
- Semaglutide (Experimental): Individuals randomized to this arm will take semaglutide once weekly.
  Interventions: Drug: Semaglutide Pen

INTERVENTIONS:
Drug: Semaglutide Pen — Individuals randomized to this arm will take semaglutide once weekly. For participants receiving in-centre hemodialysis, the intervention may be administered during the dialysis session by nursing personnel based on the patient's preference.
  Arms: Semaglutide

SUMMARY:
This study aims to determine if GLP1RA is safe and tolerable in maintenance dialysis population, adherence, and feasibility of a larger definitive cardiovascular outcome trial in this population. Participants will be randomized 1:1 to either weekly subcutaneous semaglutide versus usual care and followed for 26 weeks.

DETAILED DESCRIPTION:
In this randomized pilot study, Individuals randomized to the active intervention arm will take semaglutide once weekly. Semaglutide (injectable, 1.34 mg/mL) is delivered subcutaneously via a multiple-use pen-injector that can be used to dial in all required doses on the same pen-injector. The clinical pen has a drum scale of 1-80 in increments of 1. Participants will be trained/re-trained on injector use at 0, 4, 8, and 12 weeks. For participants receiving in-centre hemodialysis, the intervention may be administered during the dialysis session by nursing personnel. Semaglutide will be titrated using an algorithm used in previous trials with a starting dose of 0.25 mg/week, with an increase to 0.5 mg/week after 4 weeks, and to the maximum dose of 1.0 mg/week after 8 weeks as tolerated. If a participant experiences an adverse effect, efforts will be made to maintain the current dosage, with dose reductions or treatment pauses permitted at the discretion of the site investigator. Patient receiving concomitant insulin therapy will have therapy adjusted as per a pre-specified algorithm. Participants allocated to the usual care arm will receive usual care.

Primary outcomes:

1. Feasibility of study recruitment: ≥ 40% of fully eligible patients consent to participate in the trial.
2. Adherence to intervention: ≥ 70% of enrolled patients are adherent to the study intervention over the 26-week follow-up period.
3. Ability to follow: ≥ 90% of participants will be successfully followed to week

Secondary outcomes:

* Proportion Discontinuing Intervention
* Safety Events
* Major Adverse Cardiovascular Outcomes (Cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, or a peripheral arterial event)
* Body Weight/BMI
* Systolic/diastolic blood pressure
* Insulin dosage, glycemic control (HbA1c and random glucose)
* Lipid profile
* Hemoglobin, Calcium, Phosphate, PTH
* EQ-5D-5L for baseline-adjusted changes in quality of life and symptom burden

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Receiving chronic maintenance hemodialysis or peritoneal dialysis for ≥ 90 days
3. confirmed DM2 based on medical history and current or prior receipt of an oral hypoglycemic agent and/or insulin.
4. Ability to provided informed consent or through their substitute decision maker

Exclusion Criteria:

1. Type 1 DM
2. Use of a GLP-1-RA within 30 days prior to screening
3. Personal or first-degree relative(s) with a history of type 2 multiple endocrine neoplasia syndrome or medullary thyroid cancer, or acute pancreatitis (within 180 days of study screening)
4. Confirmed pregnancy, women of childbearing potential
5. Known hypersensitivity to GLP-1-RA
6. Expected to recover kidney function, stop hemodialysis, pursue palliative care, or transplantation within 6 months
7. Enrolment in another clinical trial judged by the investigator to interact with the effect of GLP1-RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adherence of Study Intervention | 26 weeks
  This will be determined if ≥ 70% of enrolled number of eligible participants (who are randomized) are adherent to the study intervention over the 26-week follow-up period.

SECONDARY OUTCOMES:
Study Medication Discontinuation | 26 weeks
  To determine the proportions of enrolled number of participants who permanently discontinue the study medication in the semaglutide arm.
Feasibility of Study Recruitment | 26 weeks
  This will be determined if ≥ 40% of the number of fully eligible participants (potential participants who were screened and identified to meet inclusion/exclusion criteria) consent to participate in the trial.
Safety Events of Special Interest | 26 weeks
  To identify safety events of special interest such as gastrointestinal symptoms, acute biliary disease, acute pancreatitis, interventions for diabetic retinopathy, heart failure exacerbations, malignant neoplasms, and the number of hypoglycemic events.
Major Adverse Cardiovascular Events | 26 weeks
  This is a composite of CV death, non-fatal myocardial infarction, non-fatal stroke, or a peripheral arterial event.
Follow Up Percentage at 26 weeks | 26 weeks
  To determine if ≥ 90% of participants (who are enrolled) will be successfully followed to week 26 (end of study participation).
Patient Reported Measures | 26 weeks
  The validated EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) score will be used to evaluate baseline-adjusted changes in quality of life and symptom burden. The EQ-5D-5L asks individuals to rate their overall health on a visual scale from 0 to 100, where 0 represents the worst imaginable health and 100 represents the best imaginable health.

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No